CLINICAL TRIAL: NCT02359435
Title: Comparison of 12-day Reverse Hybrid Therapy and 12-day Standard Triple Therapy for Helicobacter Pylori Infection - a Randomized Controlled Trial (REHYTRI Study)
Brief Title: Comparison of 12-day Reverse Hybrid Therapy and 12-day Standard Triple Therapy for Helicobacter Pylori Infection
Acronym: REHYTRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Collaborators: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KaohsiungVGH
Record Dates: First submitted 2015-01-25; First posted 2015-02-10 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Proton pump inhibitor; Eradication
MeSH Terms: interventions — Pantoprazole; Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reverse hybrid therapy (Experimental): pantoprazole 40 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg for the first 7 days, followed by pantoprazole 40 mg and amoxicillin 1 g for another 5 days; with all drugs given twice daily
  Interventions: Drug: Reverse hybrid therapy
- Standard triple therapy (Active Comparator): pantoprazole 40 mg, clarithromycin 500 mg, and amoxicillin 1 g for 12 days; with all drugs given twice daily
  Interventions: Drug: Standard triple therapy

INTERVENTIONS:
Drug: Reverse hybrid therapy — pantoprazole 40 mg b.d., amoxicillin 1 g b.d., clarithromycin 500 mg b.d. and metronidazole 500 mg b.d. for the first 7 days, followed by pantoprazole 40 mg b.d. and amoxicillin 1 g b.d. for another 5 days
  Other Names: Pantoprazole; Amoxicillin; Clarithromycin; Metronidazole
  Arms: Reverse hybrid therapy
Drug: Standard triple therapy — pantoprazole 40 mg b.d., clarithromycin 500 mg b.d., and amoxicillin 1 g b.d. for 12 days
  Other Names: Pantoprazole; Amoxicillin; Clarithromycin
  Arms: Standard triple therapy

SUMMARY:
Reverse hybrid therapy is a one-step two-phase treatment for Helicobacter pylori infection with less cost than standard triple therapy. Whether reverse hybrid therapy can replace standard triple therapy as the recommended first-line treatment is unknown. The investigators compared the efficacy of 12-day reverse hybrid therapy and 12-day standard triple therapy in first-line treatment.

DETAILED DESCRIPTION:
For this multicentre, single-blind, and randomized-controlled trial (REHYTRI study), the investigator recruited patients with H pylori infection. Using a computer-generated randomization sequence, the investigator randomly allocated patients to either 12-day reverse hybrid therapy (pantoprazole 40 mg, amoxicillin 1 g, clarithromycin 500 mg and metronidazole 500 mg for the first 7 days, followed by pantoprazole 40 mg, amoxicillin 1 g for another 5 days; with all drugs given twice daily) or a 12-day standard triple therapy (pantoprazole 40 mg, clarithromycin 500 mg, amoxicillin 1 g for 12 days; with all drugs given twice daily) at a 1:1 ratio. Our primary outcome was the eradication rate by intention-to-treat and per-protocol analyses.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H pylori-infected outpatients, at least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H pylori-eradication therapy
* ingestion of antibiotics or bismuth within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2012-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Vakil N, Megraud F. Eradication therapy for Helicobacter pylori. Gastroenterology. 2007 Sep;133(3):985-1001. doi: 10.1053/j.gastro.2007.07.008. PMID 17854602
- [Background] Hunt RH, Lam SK. Helicobacter pylori: from art to a science. J Gastroenterol Hepatol. 1998 Jan;13(1):21-8. doi: 10.1111/j.1440-1746.1998.tb00540.x. PMID 9737567
- [Background] Graham DY, Lew GM, Klein PD, Evans DG, Evans DJ Jr, Saeed ZA, Malaty HM. Effect of treatment of Helicobacter pylori infection on the long-term recurrence of gastric or duodenal ulcer. A randomized, controlled study. Ann Intern Med. 1992 May 1;116(9):705-8. doi: 10.7326/0003-4819-116-9-705. PMID 1558340
- [Background] Sung JJ, Chung SC, Ling TK, Yung MY, Leung VK, Ng EK, Li MK, Cheng AF, Li AK. Antibacterial treatment of gastric ulcers associated with Helicobacter pylori. N Engl J Med. 1995 Jan 19;332(3):139-42. doi: 10.1056/NEJM199501193320302. PMID 7800005
- [Background] Hsu PI, Lai KH, Tseng HH, Lo GH, Lo CC, Lin CK, Cheng JS, Chan HH, Ku MK, Peng NJ, Chien EJ, Chen W, Hsu PN. Eradication of Helicobacter pylori prevents ulcer development in patients with ulcer-like functional dyspepsia. Aliment Pharmacol Ther. 2001 Feb;15(2):195-201. doi: 10.1046/j.1365-2036.2001.00903.x. PMID 11148437
- [Background] Satoh K. Does eradication of Helicobacter pylori reverse atrophic gastritis or intestinal metaplasia? Data from Japan. Gastroenterol Clin North Am. 2000 Dec;29(4):829-35. doi: 10.1016/s0889-8553(05)70150-3. PMID 11190067
- [Background] Isaacson PG. Recent developments in our understanding of gastric lymphomas. Am J Surg Pathol. 1996;20 Suppl 1:S1-7. doi: 10.1097/00000478-199600001-00002. PMID 8694145
- [Background] Wong BC, Lam SK, Wong WM, Chen JS, Zheng TT, Feng RE, Lai KC, Hu WH, Yuen ST, Leung SY, Fong DY, Ho J, Ching CK, Chen JS; China Gastric Cancer Study Group. Helicobacter pylori eradication to prevent gastric cancer in a high-risk region of China: a randomized controlled trial. JAMA. 2004 Jan 14;291(2):187-94. doi: 10.1001/jama.291.2.187. PMID 14722144
- [Background] Malfertheiner P, Megraud F, O'Morain C, Bazzoli F, El-Omar E, Graham D, Hunt R, Rokkas T, Vakil N, Kuipers EJ. Current concepts in the management of Helicobacter pylori infection: the Maastricht III Consensus Report. Gut. 2007 Jun;56(6):772-81. doi: 10.1136/gut.2006.101634. Epub 2006 Dec 14. PMID 17170018
- [Background] Hsu PI, Lai KH, Lin CK, Chen WC, Yu HC, Cheng JS, Tsay FW, Wu CJ, Lo CC, Tseng HH, Yamaoka Y, Chen JL, Lo GH. A prospective randomized trial of esomeprazole- versus pantoprazole-based triple therapy for Helicobacter pylori eradication. Am J Gastroenterol. 2005 Nov;100(11):2387-92. doi: 10.1111/j.1572-0241.2005.00264.x. PMID 16279889
- [Background] Wu IC, Wu DC, Hsu PI, Lu CY, Yu FJ, Wang TE, Chang WH, Chen JJ, Kuo FC, Wu JY, Wang WM, Bair MJ. Rabeprazole- versus esomeprazole-based eradication regimens for H. pylori infection. Helicobacter. 2007 Dec;12(6):633-7. doi: 10.1111/j.1523-5378.2007.00553.x. PMID 18001406
- [Background] Fock KM, Katelaris P, Sugano K, Ang TL, Hunt R, Talley NJ, Lam SK, Xiao SD, Tan HJ, Wu CY, Jung HC, Hoang BH, Kachintorn U, Goh KL, Chiba T, Rani AA; Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol. 2009 Oct;24(10):1587-600. doi: 10.1111/j.1440-1746.2009.05982.x. PMID 19788600
- [Background] Graham DY, Fischbach L. Helicobacter pylori treatment in the era of increasing antibiotic resistance. Gut. 2010 Aug;59(8):1143-53. doi: 10.1136/gut.2009.192757. Epub 2010 Jun 4. PMID 20525969
- [Background] Graham DY, Lu H, Yamaoka Y. Therapy for Helicobacter pylori infection can be improved: sequential therapy and beyond. Drugs. 2008;68(6):725-36. doi: 10.2165/00003495-200868060-00001. PMID 18416582
- [Background] Gumurdulu Y, Serin E, Ozer B, Kayaselcuk F, Ozsahin K, Cosar AM, Gursoy M, Gur G, Yilmaz U, Boyacioglu S. Low eradication rate of Helicobacter pylori with triple 7-14 days and quadriple therapy in Turkey. World J Gastroenterol. 2004 Mar 1;10(5):668-71. doi: 10.3748/wjg.v10.i5.668. PMID 14991935
- [Background] Bigard MA, Delchier JC, Riachi G, Thibault P, Barthelemy P. One-week triple therapy using omeprazole, amoxycillin and clarithromycin for the eradication of Helicobacter pylori in patients with non-ulcer dyspepsia: influence of dosage of omeprazole and clarithromycin. Aliment Pharmacol Ther. 1998 Apr;12(4):383-8. doi: 10.1046/j.1365-2036.1998.00315.x. PMID 9690730
- [Background] Graham DY, Shiotani A. New concepts of resistance in the treatment of Helicobacter pylori infections. Nat Clin Pract Gastroenterol Hepatol. 2008 Jun;5(6):321-31. doi: 10.1038/ncpgasthep1138. Epub 2008 Apr 29. PMID 18446147
- [Background] Chuah SK, Tsay FW, Hsu PI, Wu DC. A new look at anti-Helicobacter pylori therapy. World J Gastroenterol. 2011 Sep 21;17(35):3971-5. doi: 10.3748/wjg.v17.i35.3971. PMID 22046084
- [Background] Zullo A, Vaira D, Vakil N, Hassan C, Gatta L, Ricci C, De Francesco V, Menegatti M, Tampieri A, Perna F, Rinaldi V, Perri F, Papadia C, Fornari F, Pilati S, Mete LS, Merla A, Poti R, Marinone G, Savioli A, Campo SM, Faleo D, Ierardi E, Miglioli M, Morini S. High eradication rates of Helicobacter pylori with a new sequential treatment. Aliment Pharmacol Ther. 2003 Mar 1;17(5):719-26. doi: 10.1046/j.1365-2036.2003.01461.x. PMID 12641522
- [Background] Vaira D, Zullo A, Vakil N, Gatta L, Ricci C, Perna F, Hassan C, Bernabucci V, Tampieri A, Morini S. Sequential therapy versus standard triple-drug therapy for Helicobacter pylori eradication: a randomized trial. Ann Intern Med. 2007 Apr 17;146(8):556-63. doi: 10.7326/0003-4819-146-8-200704170-00006. PMID 17438314
- [Background] Gatta L, Vakil N, Leandro G, Di Mario F, Vaira D. Sequential therapy or triple therapy for Helicobacter pylori infection: systematic review and meta-analysis of randomized controlled trials in adults and children. Am J Gastroenterol. 2009 Dec;104(12):3069-79; quiz 1080. doi: 10.1038/ajg.2009.555. Epub 2009 Oct 20. PMID 19844205
- [Background] Sanchez-Delgado J, Calvet X, Bujanda L, Gisbert JP, Tito L, Castro M. Ten-day sequential treatment for Helicobacter pylori eradication in clinical practice. Am J Gastroenterol. 2008 Sep;103(9):2220-3. doi: 10.1111/j.1572-0241.2008.01924.x. Epub 2008 Jun 28. PMID 18564109
- [Background] Tsay FW, Tseng HH, Hsu PI, Wang KM, Lee CC, Chang SN, Wang HM, Yu HC, Chen WC, Peng NJ, Lai KH, Wu DC. Sequential therapy achieves a higher eradication rate than standard triple therapy in Taiwan. J Gastroenterol Hepatol. 2012 Mar;27(3):498-503. doi: 10.1111/j.1440-1746.2011.06885.x. PMID 21871025
- [Background] Choi WH, Park DI, Oh SJ, Baek YH, Hong CH, Hong EJ, Song MJ, Park SK, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI. [Effectiveness of 10 day-sequential therapy for Helicobacter pylori eradication in Korea]. Korean J Gastroenterol. 2008 May;51(5):280-4. Korean. PMID 18516011
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Background] Greenberg ER, Anderson GL, Morgan DR, Torres J, Chey WD, Bravo LE, Dominguez RL, Ferreccio C, Herrero R, Lazcano-Ponce EC, Meza-Montenegro MM, Pena R, Pena EM, Salazar-Martinez E, Correa P, Martinez ME, Valdivieso M, Goodman GE, Crowley JJ, Baker LH. 14-day triple, 5-day concomitant, and 10-day sequential therapies for Helicobacter pylori infection in seven Latin American sites: a randomised trial. Lancet. 2011 Aug 6;378(9790):507-14. doi: 10.1016/S0140-6736(11)60825-8. Epub 2011 Jul 21. PMID 21777974
- [Background] Hsu PI, Wu DC, Wu JY, Graham DY. Modified sequential Helicobacter pylori therapy: proton pump inhibitor and amoxicillin for 14 days with clarithromycin and metronidazole added as a quadruple (hybrid) therapy for the final 7 days. Helicobacter. 2011 Apr;16(2):139-45. doi: 10.1111/j.1523-5378.2011.00828.x. PMID 21435092
- [Background] Dixon MF, Genta RM, Yardley JH, Correa P. Classification and grading of gastritis. The updated Sydney System. International Workshop on the Histopathology of Gastritis, Houston 1994. Am J Surg Pathol. 1996 Oct;20(10):1161-81. doi: 10.1097/00000478-199610000-00001. PMID 8827022
- [Background] Hsu PI, Wu DC, Chen A, Peng NJ, Tseng HH, Tsay FW, Lo GH, Lu CY, Yu FJ, Lai KH. Quadruple rescue therapy for Helicobacter pylori infection after two treatment failures. Eur J Clin Invest. 2008 Jun;38(6):404-9. doi: 10.1111/j.1365-2362.2008.01951.x. Epub 2008 Apr 22. PMID 18435764
- [Background] Kita T, Sakaeda T, Aoyama N, Sakai T, Kawahara Y, Kasuga M, Okumura K. Optimal dose of omeprazole for CYP2C19 extensive metabolizers in anti-Helicobacter pylori therapy: pharmacokinetic considerations. Biol Pharm Bull. 2002 Jul;25(7):923-7. doi: 10.1248/bpb.25.923. PMID 12132671
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1. recruitment period: Oct 2012 - Mar 2015
  2. Type of location: Kaohsiung Veterans General Hospital and Kaohsiung Medical University Chung-Ho Memorial Hospital
Pre-assignment Details: None were excluded following participant enrollment.
Period: Overall Study
Arm/Group | Reverse Hybrid Therapy | Standard Triple Therapy
Started | 220 | 220
Completed | 216 | 216
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reverse Hybrid Therapy | Standard Triple Therapy | Total
Number analyzed (Participants) | 220 | 220 | 440
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 154 | 153 | 307
  >=65 years | 66 | 67 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (12.9) | 53.4 (12.2) | 52.83 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 101 | 207
  Male | 114 | 119 | 233
Region of Enrollment [Number; unit: participants]
  Taiwan | 220 | 220 | 440

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: Evaluate eradication outcome by endoscopy urease test and histology or urea breath test
Time Frame: at the 6th week after the end of anti- H. pylori therapy
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Reverse Hybrid Therapy | Standard Triple Therapy
Number analyzed (Participants) | 220 | 220
participants | 206 | 191
Statistical Analysis 1: Comparison: Reverse Hybrid Therapy vs Standard Triple Therapy; Test type: Superiority or Other; p < 0.05, Chi-squared; Hazard Ratio (HR) = 0.016

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Reverse Hybrid Therapy | Standard Triple Therapy
Serious Adverse Events (participants affected / at risk) | 0/220 | 0/220
Other Adverse Events (participants affected / at risk) | 22/220 | 15/220
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reverse Hybrid Therapy (N=220) | Standard Triple Therapy (N=220)
Nausea (Gastrointestinal disorders) | 15 (15) | 6 (6) — Patients had Nausea discomforts.
Dizziness (Nervous system disorders) | 7 (7) | 9 (9) — Patients had dizziness discomforts.

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes